CLINICAL TRIAL: NCT05496478
Title: Assesment of Complications and Surgery Timing in Postcovid Thoracotomy Patients: Single Center Experience
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, CIGDEM YILDIRIM GUCLU, Assoc Prof Dr, Ankara University
Other Study IDs: 30250
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Thoracotomy
Keywords: Thoracotomy; covid infection; complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19 infection has caused delay in many surgeries. Besides Covid -19 infection may be a potential problem in especially major surgeries such as thoracotomies. Surgery timing, complications, intensive care unit stay and vaccination status are important issues that should be learned from post-covid cases.The aim of the study is to learn lessons from post-covid thoracotomy cases.

DETAILED DESCRIPTION:
Patients who had covid-19 infection before thoracotomy were assessed by their datas, Postoperative complications, intensive care unit stay, vaccine status, time period between covid infection and surgery were collected from patients' files and statistical analysis performed.

ELIGIBILITY:
Inclusion Criteria:

* undergoing thoracotomy
* had covid infection before surgery

Exclusion Criteria:

* age under 18
* missing data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-covid patients undergoing thoracotomy
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
number of patients who had postoperative complication | 3 days
  number of patients who had postoperative complication

CONTACTS AND LOCATIONS:
Overall Officials: CIGDEM YILDIRIM GUCLU, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No